CLINICAL TRIAL: NCT06725251
Title: The Impact of Art Therapy on the Relationships Between Individuals Diagnosed With Alzheimer's Disease and Their Care Partners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: James R. and Helen D. Russell Center for Research and Innovation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00106942; 6409 (Other: Advocate Health Care); 2016-102 (Other Grant/Funding Number: James R. and Helen D. Russell Center for Research and Innovation)
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Dementia
Keywords: self esteem; caregiver; art therapy
MeSH Terms: conditions — Dementia | interventions — Art Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dementia Participants and Care Partners (Experimental): Dyads including a participant diagnosed with dementia and the care partner
  Interventions: Behavioral: Art Therapy

INTERVENTIONS:
Behavioral: Art Therapy — Dyads will take part in a portrait-making project utilizing a collage approach. Each participant (i.e. dementia diagnosed individuals and care partners) will be instructed to create a portrait of him/herself. Participants will be provided with a sample portrait as well as bins of materials. ]The intervention will be administered for 1 ½ hours weekly, at the same day/time, for 4 consecutive weeks.

SUMMARY:
The purpose of this study is to evaluate the impact of a 4-week art therapy intervention on the relationships between individuals diagnosed with Alzheimer's disease and their care partners, on the self-esteem of diagnosed individuals, and on care partner attitudes towards persons with Alzheimer's disease.

DETAILED DESCRIPTION:
The aim is to develop and implement an art therapy intervention for dyads - each consisting of an individual diagnosed with mild Alzheimer's disease and his/her care partner - with the goals of improving patients' and care partners' sense of their relationship, increasing patients' self-esteem and improving care partner attitudes towards individuals with Alzheimer's disease. The specific intervention will be a portrait-making project utilizing a collage approach. Each participant (i.e. diagnosed individuals and care partners) will be instructed to create a portrait of him/herself. Participants will be provided with a sample portrait as well as bins of materials (e.g. words, images, markers). The intervention will be administered for 1 ½ hours weekly, at the same day/time, for 4 consecutive weeks.

ELIGIBILITY:
Inclusion criteria for patients include:

* A diagnosis of Alzheimer's disease, based on the NIA/AA Diagnostic Guidelines for Alzheimer's Disease (McKhann et al., 2011)
* MMSE of 18-26, inclusive, administered within 6 month prior to screening or at screening
* Awareness of diagnosis and/or memory impairment, as determined by semi-structured interview with clinician (see Appendix B)
* Availability and willingness to participate in all 4 sessions of the intervention
* A care partner with whom the patient has regular weekly contact and who is available and willing to participate in all 4 sessions of the intervention
* Sufficient visual acuity to read 12-point font
* Sufficient manual dexterity to use scissors
* Ability to hear instructions in a classroom setting
* Ability to read English
* Age 18 years old or greater

Exclusion criteria for patients include:

* Any uncontrolled medical or neurological/neurodegenerative condition (other than AD) that, in the opinion of the Investigator, might be a contributing cause of the subject's cognitive impairment (e.g., substance abuse, vitamin B12 deficiency, abnormal thyroid function, stroke or other cerebrovascular condition, Lewy body dementia, fronto-temporal dementia, head trauma).
* Current active psychiatric illness (e.g., major depression, schizophrenia, etc.)
* Current active seizure disorder.
* Malignancy or carcinoma currently requiring active treatment or progressing off of treatment.
* Recent history (within 1 year) of alcohol abuse or drug abuse.
* Active tobacco use that interferes with visits (e.g., if the patient would need to smoke during the therapy session).
* Use of medications (e.g., narcotics, sedatives, etc.) that lead to drowsiness during the therapy sessions
* Inability to comply with the instructions of the art therapist.
* Other unspecified reasons that, in the opinion of the Investigator make the subject unsuitable for enrollment.
* Prisoners

Inclusion criteria for care partners include:

* Adult 18 years of age or older
* Ability to consent
* Regular weekly contact with the subject diagnosed with Alzheimer's disease
* Availability and willingness to participate in all 4 sessions of the intervention
* Sufficient visual acuity to read 12-point font
* Sufficient manual dexterity to use scissors
* Ability to hear instructions in a classroom setting
* Ability to read English

Exclusion criteria for care partners include:

* Any uncontrolled medical or neurological/neurodegenerative condition sufficient to cause cognitive impairment
* Current active psychiatric illness (e.g., major depression, schizophrenia, etc.)
* Current active seizure disorder.
* Malignancy or carcinoma currently requiring active treatment or progressing off of treatment.
* Recent history (within 1 year) of alcohol abuse or drug abuse.
* Active tobacco use that interferes with visits (e.g., if the care partner would need to smoke during the therapy session).

Use of medications (e.g., narcotics, sedatives, etc.) that lead to drowsiness during the therapy sessions

* Inability to comply with the instructions of the art therapist.
* Other unspecified reasons that, in the opinion of the Investigator make the care partner unsuitable for enrollment.
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-08-26 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-08-02 (Actual)

PRIMARY OUTCOMES:
Impact of Art Therapy on Quality of Dyadic Relationship | Week 1
  Impact of art therapy on quality of dyadic relationship will be determined using the Dyadic Relationship Scale. The survey consists of 10 questions with a total score range of 10-40. The score is a measure of patient and care partner perceptions of their relationship. Lower scores indicate the perception of a poorer relationship (i.e. greater strain, lower positive interactions) and higher scores indicate a perceived better relationship (i.e. lower strain, greater positive interactions).
Impact of Art Therapy on Quality of Dyadic Relationship | Week 4
  Impact of art therapy on quality of dyadic relationship will be determined using the Dyadic Relationship Scale. The survey consists of 10 questions with a total score range of 10-40. The score is a measure of patient and care partner perceptions of their relationship. Lower scores indicate the perception of a poorer relationship (i.e. greater strain, lower positive interactions) and higher scores indicate a perceived better relationship (i.e. lower strain, greater positive interactions).

SECONDARY OUTCOMES:
Impact of Art Therapy on Dementia Individuals' Self-esteem | Week 1
  The impact of art therapy on the dementia diagnosed individuals' self-esteem will be determined by the Rosenberg Self-Esteem Scale. The survey consists of 10 questions with a total score range of 0-30. The score is a measure of patient self-esteem, with lower scores meaning lower self-esteem and higher scores meaning higher self-esteem.
Impact of Art Therapy on Dementia Individuals' Self-esteem | Week 4
  The impact of art therapy on the dementia diagnosed individuals' self-esteem will be determined by the Rosenberg Self-Esteem Scale. The survey consists of 10 questions with a total score range of 0-30. The score is a measure of patient self-esteem, with lower scores meaning lower self-esteem and higher scores meaning higher self-esteem.
Impact of Art Therapy on Dementia Individuals' Sense of Stigma | Week 1
  The impact of art therapy on diagnosed individuals' sense of stigma will be determined by the Stigma Impact Scale. The survey consists of 20 questions with a total score range of 0-80. The score is a measure of the patient's perception of stigma, with lower scores indicating lower perceived stigma and higher scores indicating greater perceived stigma.
Impact of Art Therapy on Dementia Individuals' Sense of Stigma | Week 4
  The impact of art therapy on diagnosed individuals' sense of stigma will be determined by the Stigma Impact Scale. The survey consists of 20 questions with a total score range of 0-80. The score is a measure of the patient's perception of stigma, with lower scores indicating lower perceived stigma and higher scores indicating greater perceived stigma.
Impact of Art Therapy on Care Partner Attitudes Towards Persons with Dementia | Week 1
  The impact of art therapy on care partner attitudes towards persons with dementia will be determined by the Dementia Attitudes Scale. The survey consists of 20 questions with a total score range of 20-140. The score is a measure of care partner attitudes towards patients with dementia. Lower scores indicate lower knowledge and social comfort with persons with dementia and a higher score indicates greater knowledge and social comfort with persons with dementia.
Impact of Art Therapy on Care Partner Attitudes Towards Persons with Dementia | Week 4
  The impact of art therapy on care partner attitudes towards persons with dementia will be determined by the Dementia Attitudes Scale. The survey consists of 20 questions with a total score range of 20-140. The score is a measure of care partner attitudes towards patients with dementia. Lower scores indicate lower knowledge and social comfort with persons with dementia and a higher score indicates greater knowledge and social comfort with persons with dementia.

CONTACTS AND LOCATIONS:
Overall Officials: Darren Gitelman, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Advocate Memory Center, Park Ridge, Illinois, United States

IPD SHARING:
Plan to Share IPD: No